CLINICAL TRIAL: NCT02984878
Title: A Multicenter, Double-Blind, Randomized, Split-Face Study to Evaluate the Safety and Efficacy of Revanesse® Ultra (Retreatment)
Brief Title: Multicenter Study to Evaluate the Safety and Efficacy of Revanesse® Ultra Retreatment
Acronym: Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prollenium Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYM2014-02 Retreatment
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-10

CONDITIONS: Nasolabial Fold Correction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Revanesse Ultra (Experimental): Revanesse Ultra open label retreatment
  Interventions: Device: Revanesse Ultra

INTERVENTIONS:
Device: Revanesse Ultra — Nasolabial Fold correction

SUMMARY:
To compare improvement with retreatment for all subjects undergoing correction of nasolabial folds (NLFs) in the initial SYM2014-02 study, who were retreated with Revanesse Ultra at Visit 6/Week 24 and to determine the safety of repeat injections of Revanesse Ultra. The retreatment phase was optional.

DETAILED DESCRIPTION:
The subjects completing the initial phase of the SYM2014-02 study (NCT02987205) who had returned to baseline Wrinkle Severity Rating Scale (WSRS) score or as needed for optimal correction if WSRS scores had not returned to baseline, were offered the option for retreatment with Revanesse Ultra

Visit 6/Week 24 (± 7 days) optional open-label retreatment with Revanesse Ultra for subjects who had returned to baseline Wrinkle Severity Rating Scale (WSRS) score or as needed for optimal correction if WSRS scores had not returned to baseline; End of Study for subjects not being retreated

Visit 7/Week 28 (± 7 days) follow-up for retreated subjects

Visit 8/Week 52 (± 7 days) End of Study for retreated subjects

A telephone contact was performed at Week 40 (± 7 days) for retreated subjects to assess adverse events (AEs) and concomitant medications.

This report presents the results for all subjects who received optional open-label retreatment with Revanesse Ultra at Visit 6/Week 24.

This study was performed in compliance with Good Clinical Practice (GCP), including the archiving of essential documents.

Number of Subjects (Planned and Analyzed): Seventy-one subjects received retreatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects from the SYM2014-02 initial study who were:

* Men or women at least 22 years of age with two fully visible bilateral nasolabial folds each with a WSRS score of 3 or 4 (moderate or severe) that may have been corrected with an injectable dermal filler.
* Subjects were eligible for retreatment when WSRS scores had returned to baseline for either or both NLFs (retreatment group).
* If scores had not returned to baseline, subjects were also eligible to be injected for either one or both NLFs as needed to achieve optimal correction (optimal correction group).

Exclusion Criteria:

-

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Gold, MD, Principal Investigator — Tennessee Clinical Research Center

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Revanesse Ultra Retreatment: Revanesse Ultra: Nasolabial Fold correction - - Subjects could have open-label retreatment as needed with Revanesse Ultra at 6 months if their WSRS scores had returned to baseline
- Revanesse Ultra Optimal Correction: The Optimal Correction group scores had not returned to baseline, subjects were eligible to be injected for either one or both NLFs as needed to achieve optimal correction (optimal correction group).
Period: Overall Study
Arm/Group | Revanesse Ultra Retreatment | Revanesse Ultra Optimal Correction
Started | 30 | 41
Completed | 30 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Revanesse Ultra open label retreatment / Nasolabial Fold correction - optional open-label retreatment with Revanesse Ultra for subjects who had returned to baseline Wrinkle Severity Rating Scale (WSRS) score or as needed for optimal correction if WSRS scores had not returned to baseline.
Groups:
- Revanesse Ultra Retreatment: Revanesse Ultra open label retreatment / Nasolabial Fold correction - optional open-label retreatment with Revanesse Ultra for subjects who had returned to baseline Wrinkle Severity Rating Scale (WSRS) score The subjects completing the initial phase of the SYM2014-02 study (NCT02987205) who had returned to baseline Wrinkle Severity Rating Scale (WSRS) score, were offered the option for retreatment with Revanesse Ultra Safety data was collected to assess treatment emergent adverse events associated with repeat injections. Seventy-one subjects received retreatment - 30 returned to baseline
- Revanesse Ultra Optimal Correction: Revanesse Ultra open label retreatment / Nasolabial Fold correction - optional open-label retreatment with Revanesse Ultra for subjects as needed for optimal correction if WSRS scores had not returned to baseline.
  The subjects completing the initial phase of the SYM2014-02 study (NCT02987205) were treated as needed for optimal correction if WSRS scores had not returned to baseline, and were offered the option for retreatment with Revanesse Ultra Safety data was collected to assess treatment emergent adverse events associated with repeat injections. Seventy-one subjects received retreatment - 41 were included in the optimal correction group
- Total: Total of all reporting groups
Arm/Group | Revanesse Ultra Retreatment | Revanesse Ultra Optimal Correction | Total
Number analyzed (Participants) | 30 | 41 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (9.19) | 54.5 (10.44) | 56.1 (10.05)
Age, Customized [Count of Participants; unit: Participants] — participants in each age group
  Participants
    22 to <40 years | 1 | 5 | 6
    40 to <64 years | 21 | 27 | 48
    64 to <75 years | 6 | 9 | 15
    > = 75 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 37 | 66
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 26 | 33 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 29 | 37 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 41 | 71
Fitzpatrick Skin Type (FST) Classification [Count of Participants; unit: Participants] — FST Type I skin always burns, never tans (pale white; blond or red hair; blue, gray eyes; freckles), FST Type II skin usually burns, tans minimally (white; blond, brown or red hair; blue, green, or hazel eyes), FST Type III skin sometimes has a mild burn, tans uniformly (cream white; yellowish; any hair color or brown eyes), FST Type IV skin burns minimally, always tans well (light brown; olive; dark brown to black hair), FST Type V skin very rarely burns, tans very easily (brown), FST Type VI skin never burns, always tans (deeply pigmented dark brown to darkest brown, black in complexion)
  Participants
    FST I | 0 | 0 | 0
    FST II | 10 | 17 | 27
    FST III | 15 | 15 | 30
    FST IV | 3 | 3 | 6
    FST V | 1 | 2 | 3
    FST VI | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in the Wrinkle Severity Rating Scale (WSRS) With Subjects From Both the Retreatment and the Optimal Correction Groups - WSRS Scores at Visit 8/Week 52
Description: Change in the Wrinkle Severity Rating Scale (WSRS) With Subjects From Both the Retreatment and the Optimal Correction Groups Achieving Similar WSRS Scores at Visit 8/Week 52 - WSRS Score categories: 1. Absent - No visible fold; continuous skin line. 2. Mild - Shallow but visible fold with a slight indentation; minor facial feature; implant is expected to produce a slight improvement in appearance. 3. Moderate - Moderately deep folds; clear facial feature visible at normal appearance but not when stretched; excellent correction is expected from injectable implant. 4. Severe - Very long and deep folds; prominent facial feature; less than 2 mm visible when stretched; significant improvement is expected from injectable implant. 5. Extreme - Extremely deep and long folds, detrimental to facial appearance; 2 to 4 mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone. An increase in the WSRS score indicates a worsening of severity.
Time Frame: Visit 8/Week 52
Population: Subjects that completed the SYM 2014-02 Main Study were eligible for the SYM 2014-02 Retreatment Study.
Measure: Mean (Standard Deviation); unit: units on WSRS scale
Units Other Than Participants: Nasolabial Folds
Groups:
- Optimal Correction Group: Optional Open label Retreatment at Week 24 / SYM2014-02 Retreatment: At SYM 2014-02 Main Study Visit 6/Week 24, a subject could be retreated with Revanesse Ultra. Subjects were eligible for optimal correction when WSRS scores had not returned to baseline. Optimal Correction subjects were injected in either one or both NLFs as needed to achieve optimal correction. These subjects continued to day 196 (Visit 7 / week 28), received a phone contact at day 280 (week 40), and completed at day 364 (Visit 8 / week 52).
- Retreatment Group: Revanesse Ultra open label retreatment for Nasolabial Fold correction. Optional Open-label Retreatment at Visit 6/Week 24 of the SYM 2014-02 Main Study, a subject could be retreated when WSRS scores had returned to baseline for either or both NLFs. The retreatment group and the optimal correction group were separated for data analysis. These subjects continued to day 196 (Visit 7 / week 28), received a phone contact at day 280 (week 40), and completed at day 364 (Visit 8 / week 52).
Arm/Group | Optimal Correction Group | Retreatment Group
Number analyzed (Participants) | 41 | 30
Number analyzed (Nasolabial Folds) | 81 | 60
units on WSRS scale
  Change in Main Study Treatment - Revanesse Ultra | 0.1 (0.69) | 0.6 (0.72)
  Change in Main Study Treatment - Restylane | 0.0 (0.69) | 0.8 (0.63)

2. Secondary Outcome: Retreatment Safety Assessed by the Incidence of Adverse Events (AEs), Which Were Defined, Recorded, Reported, and Evaluated, by Number and Severity
Description: Assess safety concerns with retreatment of Revanesse Ultra for men or women at least 22 years of age with NLFs with a moderate or severe WSRS score at baseline who had previously received 1 or 2 treatments with Restylane or Revanesse Ultra, Adverse Events (AEs), which were defined, recorded, reported, and evaluated
Time Frame: Visit 6/Week 24, Visit 7/Week 28, Visit 8/Week 52
Population: Counts reflect numbers of subjects reporting one or more injection site TEAE that map to the MedDRA (version 15.1) system organ class/preferred term. At each level of summarization (system organ class or preferred term), subjects reporting more than one injection site TEAE are counted only once.
Measure: Count of Participants; unit: Participants
Arm/Group | Revanesse Ultra Retreatment | Revanesse Ultra Optimal Correction
Number analyzed (Participants) | 30 | 41
Participants
  Eye disorder - ocular hyperaemia | 0 | 1
  Gastrointestinal - mouth cyst | 0 | 1
  Injection site erythema | 2 | 8
  Injection site haematoma | 9 | 19
  Injection site mass | 1 | 2
  Injection site pain | 9 | 6
  Injection site pruritis | 0 | 1
  Injection site swelling | 0 | 1
  Contusion | 0 | 1
  Excoriation | 0 | 1

3. Secondary Outcome: Patient Global Aesthetic Improvement (pGAI) Score
Description: Subjects were evaluated on the Patient Global Aesthetic Improvement (pGAI) Patient Global Aesthetic Improvement (pGAI) Score: 1 = Worse, 2 = No change, 3 = Improved, 4 = Much improved, 5 = Very much improved
Time Frame: Visit 8/Week 52
Population: Subjects were evaluated on the Patient Global Aesthetic Improvement (pGAI)
Measure: Count of Participants; unit: Participants
Groups:
- Revanesse Ultra Retreatment: Revanesse Ultra: Nasolabial Fold correction - Subjects could have open-label retreatment as needed with Revanesse Ultra at 6 months if their WSRS scores had returned to baseline
Arm/Group | Revanesse Ultra Retreatment | Revanesse Ultra Optimal Correction
Number analyzed (Participants) | 30 | 41
Participants
  Visit 8 - week 52 pGAI = 1 worse | 1 | 1
  Visit 8 - week 52 pGAI = 2 no change | 8 | 8
  Visit 8 - week 52 pGAI = 3 Improved | 13 | 16
  Visit 8 - week 52 pGAI = 4 much improved | 1 | 12
  Visit 8 - week 52 pGAI = 5 Very much improved | 7 | 4

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected at Retreatment for 6 months (Visit 8/Week 52 from the Main Study)
Description: Treatment safety was evaluated by frequency and percent of subjects and investigators reporting treatment-emergent adverse events (TEAEs) tabulated by treatment group, location, frequency, severity and duration after each treatment (initial treatment, touch up) and throughout the study. TEAEs were assessed by a subject diary after each injection, touch up and follow up visit, and were reported by the Evaluating Investigator at each of the follow-up visits.
Arm/Group | Retreatment Group | Optimal Correction Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/41
Other Adverse Events (participants affected / at risk) | 16/30 | 29/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Retreatment Group (N=30) | Optimal Correction Group (N=41)
INJECTION SITE ERYTHEMA (General disorders) | 2 (2) | 9 (9) — Counts reflect numbers of subjects reporting one or more injection site TEAEs that map to the MedDRA (version 15.1). At each level of summarization (SOC or preferred term) subjects reporting more than one injection site TEAE are only counted once.
INJECTION SITE HAEMATOMA (General disorders) | 9 (9) | 19 (19) — bruising
INJECTION SITE PAIN (General disorders) | 9 (9) | 6 (6) — pain at the injection site
INJECTION SITE SWELLING (General disorders) | 9 (9) | 14 (14) — Swelling at the injection site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions within the site contracts, sites cannot publish any results and also have confidentiality agreements in place separately that restrict any publications by sites regarding results, findings, etc.

DOCUMENTS (1):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT02984878/Prot_000.pdf